CLINICAL TRIAL: NCT05012059
Title: A Comparison of General Versus Peripheral Nerve Block for Lower Extremity Amputation in Diabetic Patients With Bleeding Tendency: a Retrospective Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2021-0378
Record Dates: First submitted 2021-08-16; First posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Daibetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective data collection. The aim of this study is to compare general anesthesia and nerve block anesthesia with respect to the postoperative complications in patients undergoing diabetic leg amputation and having bleeding tendency.

ELIGIBILITY:
Inclusion Criteria:

1.Adults patients ≥20 years who underwent lower extremity amputation for diabetic foot under general anesthesia or PNB and having coagulopathy in which condition that neuraxial block is contraindicated

Exclusion Criteria:

1. patients with prior surgical history within 1 month
2. combined operation (joint operation)
3. patients who required continuous intravenous administration of vasopressors and/or mechanical ventilation prior to surgery
4. combination of general anesthesia and PNB

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients ≥20 years who underwent lower extremity amputation for diabetic foot under general anesthesia or PNB and having coagulopathy in which condition that neuraxial block is contraindicated
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Occurrence of major complication | Within 1 month after the surgery
  Major complications included pneumonia (followed the definition of European Perioperative Clinical Outcome), myocardial infarction (followed the definition of World Health Organization), stroke (A central neurologic deficit persisting postoperatively for > 24 h), venous thromboembolism (confirmed by image study), delirium (confirmed by psychiatrist), acute kidney injury (based on Kidney Disease: Improving Global Outcomes Criteria), new requirement for dialysis, surgical site infection, Return to the OP room.
Occurrence of mortality | Within 1 month after the surgery
  Mortality refers all deaths.

CONTACTS AND LOCATIONS:
Overall Officials: Hye Jin Kim, Principal Investigator — Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided